CLINICAL TRIAL: NCT06090799
Title: A Study of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SHR-3032 Following Single Intravenous Administration in Healthy Subjects
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SHR-3032 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong Hengrui Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-3032-101
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Prevention of Graft Rejection After Organ Transplantation

STUDY DESIGN:
Intervention Model Description: SHR-3032 for dose escalation
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A (Experimental): SHR-3032
  Interventions: Drug: SHR-3032
- Treatment group B (Placebo Comparator): SHR-3032 Placebo
  Interventions: Drug: SHR-3032 Placebo

INTERVENTIONS:
Drug: SHR-3032 — Single dose at varying dosage levels depending on treatment assignment
  Arms: Treatment group A
Drug: SHR-3032 Placebo — Single dose at varying dosage levels depending on treatment assignment
  Arms: Treatment group B

SUMMARY:
This is a single-center, double-blind, dose-escalation study to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of SHR-3032 in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

1. The age when signing the informed consent form is between 18 and 55 years old (inclusive);
2. Male weight ≥ 50 kg and female weight ≥ 45 kg, body mass index (BMI) is between 19.0 ~ 28.0 kg/m2 (inclusive) during the screening period;
3. The subject has no plans to donate sperm or eggs from signing the informed consent form to 6 months following administration. Female subjects with reproductive potential must conduct a serum pregnancy test within 7 days before the first drug use, and the result is Negative. Fertile female subjects and male subjects whose partners are females of childbearing age must agree to comply with contraceptive requirements from signing the informed consent form to 6 months following administration;
4. Female subjects: non-pregnant or non-lactating;
5. The subject has a detailed understanding of the nature, significance, possible benefits, possible inconvenience, potential risks and discomfort of the study, can understand the procedures and methods of this study, and is willing to strictly abide by the requirements of the entire clinical study and voluntarily signed the informed consent.

Exclusion Criteria:

1. Previously or currently suffering from clinical acute and chronic diseases of circulatory system, endocrine system, nervous system, digestive system, respiratory system, hematology, immunology, psychiatry and metabolic abnormalities, who are judged by the researchers to be inappropriate for enrollment;
2. During the screening period, aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥ 2 times the upper limit of the normal range (ULN), or total bilirubin (TBIL) ≥ 1.5 times the ULN, or lymphocytes were lower than the lower limit of the normal range;
3. The subjects' medical history, symptoms and examination results at the time of screening suggest that they have active tuberculosis or latent tuberculosis;
4. Those who had chronic infection or recurrent infection and needed treatment within 12 months before screening;
5. People with hereditary bleeding or coagulation disorders, or a history of non-traumatic bleeding (bleeding requiring treatment);
6. Those who are at risk of thromboembolic events (such as thromboembolism in cardiovascular, cerebrovascular, peripheral blood vessels);
7. Previous medical history of torsade de pointes, symptomatic ventricular arrhythmia, or personal or family history of short QT syndrome or long QT syndrome;
8. Patients with abnormal and clinically significant hyperkalemia and hypokalemia judged by the investigator;
9. People who are known to have a history of allergies to this product, its excipients, similar drugs, or allergic constitution (allergic to 2 or more drugs and food);
10. Those who have undergone major surgery within 3 months before screening, or those who have previously received surgery that may significantly affect the pharmacokinetic characteristics or safety evaluation of the investigational drug, or those who plan to undergo surgery during the study period;
11. Any drug that inhibits or induces liver metabolism of drug has been used within 1 month before administration (such as: inducers-barbiturates, carbamazepine, phenytoin, glucocorticoids, omeprazole; inhibitors- SSRI antidepressants, cimetidine, diltiazem, macrolides, nitroimidazoles, sedative hypnotics, verapamil, fluoroquinolones, antihistamines);
12. Those who have been vaccinated within 1 month before screening or plan to be vaccinated during the study;
13. Those who have used any drugs or health products (including Chinese herbal medicines) within 7 half-lives or 14 days (whichever is longer) before the administration, or those who are known during the screening period may need to receive other drug treatments during the study;
14. Those who have participated in clinical trials and received experimental drugs within 3 months before screening, or plan to participate in other clinical trials during this study;
15. Those who have received any systemic glucocorticoid therapy within 3 months before screening;
16. Those who have received any of the following treatments at any time before: B cell targeted therapy; Abatacept;
17. Donate blood/blood loss ≥ 400 mL within 3 months before screening (except for female physiological blood loss), receive blood transfusion or use blood products, or plan to donate blood during the test or within 1 month after the end of the test;
18. Those who smoked more than 5 cigarettes per day on average within 3 months before screening, or who could not quit smoking during the study;
19. Regular drinkers within 3 months before screening (drinking more than 14 units of alcohol per week on average, 1 unit = 360 mL of beer or 45 mL of 40% spirits or 150 mL of wine), or unable to stop drinking during the study;
20. Those who drank excessive tea, coffee or caffeinated beverages (average of more than 8 cups per day, 1 cup = 200 mL) within 3 months before screening;
21. Those who consumed special food (such as grapefruit, grapefruit juice or food/drink containing grapefruit juice, chocolate, tobacco, alcohol, caffeine and other food or drink) within 48 hours before administration;
22. Those who have special requirements for diet and cannot follow a unified diet;
23. Screening period or baseline examination results (vital signs, physical examination, 12-lead electrocardiogram, lateral chest X-ray, abdominal B-ultrasound, thyroid function, blood routine, urine routine, stool routine, blood biochemistry, coagulation function test) are abnormal and have clinical significance judged by the investigators;
24. One or more positive tests for hepatitis B surface antigen, hepatitis C virus antibody, syphilis or human immunodeficiency virus antibody;
25. Those who have a history of drug abuse or who are positive for drug abuse screening;
26. Alcohol breath screening results are positive;
27. Those who have difficulty in venous blood collection or who cannot tolerate venipuncture, or those who have a history of fainting of needles and blood;
28. The subject may not be able to complete the study due to other reasons or the investigators considers that he is not suitable for inclusion.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2023-11-29 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-04-08 (Actual)

PRIMARY OUTCOMES:
The incidence and severity of adverse events/serious adverse events | From ICF signing date to day 99
Pharmacokinetic parameter of SHR-3032: Cmax | 0 minute to day 99 after administration
Pharmacokinetic parameter of SHR-3032: AUC0-t | 0 minute to day 99 after administration
Pharmacokinetic parameter of SHR-3032: AUC0-∞ | 0 minute to day 99 after administration
Pharmacokinetic parameter of SHR-3032: Tmax | 0 minute to day 99 after administration
Pharmacokinetic parameter of SHR-3032: t1/2 | 0 minute to day 99 after administration
Pharmacokinetic parameter of SHR-3032: CL | 0 minute to day 99 after administration
Pharmacokinetic parameter of SHR-3032: Vss | 0 minute to day 99 after administration

SECONDARY OUTCOMES:
The percentage of target receptor occupancy | 0 minute to day 99 after administration
The incidence of positive ADA | 0 minute to day 99 after administration

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided